CLINICAL TRIAL: NCT04207619
Title: Evaluating Glial Acetate Metabolism as a Biomarker of Hypoglycemic Counterregulation Using 13C Magnetic Resonance Spectroscopy.
Brief Title: Evaluating Glial Acetate Metabolism as a Biomarker of Hypoglycemic Counterregulation
Acronym: E-VAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, David McDougal, Assistant Professor, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBRC 2019-047
Record Dates: First submitted 2019-12-17; First posted 2019-12-23 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Diabetes; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Participants will have their glial acetate metabolism measured by carbon-13 magnetic resonance spectroscopy as well as their neuroendocrine response to hypoglycemia 3 days later.
  Interventions: Other: hyperinsulinemic-hypoglycemic clamp; Other: 13C-MRS procedure/Acetate infusion

INTERVENTIONS:
Other: hyperinsulinemic-hypoglycemic clamp — An intravenous catheter will be placed in an antecubital vein for infusion of insulin and glucose. A second catheter will be placed retrograde in a dorsal vein of the contra-lateral hand for blood withdrawal. The hand will be placed in a heating box or pad at 70°C for arterialization of venous blood. A primed infusion of regular insulin (120 mU/min/m2) will be initiated and continued for approximately 2 hours. Beginning 20 minutes prior to the start of the insulin infusion, arterialized venous blood glucose will be measured at 5 minute intervals via a Hemocue or YSI analyzer. Following initiation of insulin infusion, blood glucose will be allowed to fall to 50 mg/dL and then maintained at this level using a variable infusion of exogenous dextrose (20% solution). Our goal is to achieve steady-state (blood glucose stabilized at 50 +/- 5 mg/dL) within the first 45 minutes following the start of insulin infusion.
Other: 13C-MRS procedure/Acetate infusion — Glial metabolism will be measured via MRS utilizing a simultaneous intravenous infusion of 13C labeled acetate. An intravenous catheter will be placed in a vein of each arm, one to infuse 13C-acetate and the other to draw blood samples

SUMMARY:
Hypoglycemic complications are a major impediment to the maintenance of healthy glucose levels in persons with diabetes. The investigators recently completed a clinical pilot and feasibility study (GLIMPSE, NCT02690168), which identified a novel biomarker, glial acetate metabolism, that appears to predict the susceptibility to hypoglycemia. By providing an assay to predict hypoglycemic events and therefore diabetic complications, the development of this biomarker could significantly improve the treatment of persons with diabetes.

The goal of this study is to determine the efficacy of our biomarker for predicting susceptibility to insulin-induced hypoglycemia. In order to accomplish this goal the investigatiors will pair our 13C magnetic resonance spectroscopy procedure to assess glial acetate metabolism, developed in the GLIMPSE study, with a hyperinsulinemic-hypoglycemic clamp procedure, developed in the HYPOCLAMP study (NCT03839511). The two procedures will be separated by a three day interval. The investigators will then correlate the participants' rates of glial acetate metabolism with their neuroendocrine responses to the hypoglycemic clamp. This proof of concept study will test the hypothesis that glial acetate metabolism is inversely proportional to the neuroendocrine response to hypoglycemia, that is, as glial acetate metabolism increases the neuroendocrine response will decrease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Ages 18-40 years
* BMI between 20 kg/m2 and 30 kg/m2 (±0.5 kg/m2 will be accepted)
* Medically cleared for participation in the study

Exclusion Criteria:

* Contraindication to MRI
* Consume >10 alcoholic drinks/week
* History of chronic smoking or have quit less than 10 years ago
* History of clinically diagnosed diabetes or a fasting blood glucose >126 mg/dL
* Average screening blood pressure >140/90 mmHg
* History of cardiovascular disease
* Pregnant, planning to become pregnant, or breastfeeding
* Use of medications affecting glucose metabolism, e.g., benzodiazepines, thiazide diuretics, cortisone, and prednisone.
* Use of beta-adrenergic antagonists.
* Based on the investigative team's clinical judgement, a subject may not be appropriate for participation in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent 13C enrichment of bicarbonate measured via carbon-13 magnetic resonance spectroscopy (13C-MRS) | Every ten minutes for 120 minutes following administration of 1-13C acetate
  Glial acetate metabolism

SECONDARY OUTCOMES:
Change in serum epinephrine levels | epinephrine will be measured every 15 minutes for 135 minutes.
  The change is serum epinephrine during the hypoglycemic clamp will be determined relative to baseline levels

CONTACTS AND LOCATIONS:
Overall Officials: David McDougal, PhD, Principal Investigator — PBRC
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No